CLINICAL TRIAL: NCT03109444
Title: Normative Radiographic Parameters and Growth Curve of Hips Less Than Six Weeks of Gestational Age Using Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: Hip Growth Chart
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Newborn; Hip Dysplasia
Keywords: Hip Growth Chart
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip Ultrasound of Newborn infants: Newborns born at CRMC (term newborns and pre-mature newborns over 32 weeks gestational age). This will include newborns cared for in the neonatal intensive care unit (NICU) over 32 weeks gestational age, and newborns cared for on the normal labor and delivery floor. the newborn will receive an ultrasound of their hips while in the hospital (done by a trained sonographer). This will happen in the patient's room with the LAR present. An ultrasound of the hip takes approximately 15 minutes and is non-invasive, non-painful and does not utilize any ionizing radiation. Newborns will be scheduled to return once a week until the newborn's hips reach criteria for normal hip morphology or the newborn reaches 6 weeks of corrected age.
  Interventions: Diagnostic Test: Hip Ultrasound

INTERVENTIONS:
Diagnostic Test: Hip Ultrasound — Both hips will be examined. The diagnostic examination for developmental dysplasia of the hip (DDH) incorporates 2 orthogonal planes: a coronal view in the standard plane at rest and a transverse view of the flexed hip at rest. It is acceptable to perform the examination with the infant in a supine or a lateral decubitus position. The anatomic coronal plane is approximately parallel to the posterior skin surface of an infant. The imaging plane is through the deepest part of the acetabulum (which includes visualization of the triradiate cartilage and the ischium posteriorly), the resulting image will be a coronal view in the standard plane. The standard plane is defined by identifying a straight iliac line, the tip of the acetabular labrum, and the transition from the os ilium to the triradiate cartilage. Acetabular morphology is assessed in this view and may be validated by measuring the acetabular alpha angle (≥60°). The femoral head coverage by the bony acetabulum should be >50%.

SUMMARY:
This study aims to collect normative population data on the ultrasound radiographic parameters used to evaluate hip dysplasia in infants between 32 and 46 weeks of gestational age. This data would be utilized to develop a growth chart with standard deviations for this cohort that would be beneficial in the appropriate treatment of suspected hip dysplasia.

DETAILED DESCRIPTION:
This is a prospective population cohort study of newborns that are born at Community Regional Medical Center (CRMC). Legally authorized representatives (LAR) of the newborn will be approached by research staff after the birth of their baby, informed about the study and then asked if they would like to participate. Due to the high volume of births at CRMC, LARs will be approached approximately once a week for a convenience sample.

If a LAR is interested in participating, they will be consented to be in the study.

After a LAR consents for participation the newborn will receive an ultrasound of their hips while in the hospital (done by a trained sonographer). This will happen in the patient's room with the LAR present. An ultrasound of the hip takes approximately 15 minutes and is non-invasive, non-painful and does not utilize any ionizing radiation.

Study Follow-Up LARs and newborns will be scheduled to return once a week until the newborn's hips reach criteria for normal hip morphology or the newborn reaches 6 weeks of corrected age. Normal infant hip ultrasound maturity is defined as an alpha angle of > 60 degrees (this is the angle between the roof of the acetabulum and the lateral iliac wing and indicates morphology of the acetabulum) and a percent coverage of the femoral head in the acetabulum of > 50%. A Board Certified Pediatric Radiologist, a Board Certified Pediatric Orthopaedic Surgeon and an Orthopaedic Resident will interpret each study. If there is less than 5 degree or 5 percent difference between the interpretations the mean will be used as the reading. If there is a greater difference, the case will be reviewed for consensus. Corrected age is defined as actual age in weeks minus weeks premature. For example, a newborn born at 32 weeks gestational age (8 weeks premature) would be followed for 14 weeks total (14 weeks actual age-8 weeks premature=6 weeks adjusted age).

If a newborns hips reach the criteria for newborn hips before they reach 6 weeks adjusted age, they will discharged from the study as they have reached the standard for infant hip maturity (this could happen at their initial scan or any time after). LAR and newborns will return to CRMC Radiology Department to get the follow up ultrasounds therefore there will be an incentive of $15 a follow up visit. Incentive will not be provided for studies performed while a hospital inpatient. If a patient shows persistent radiographic signs of dysplasia at any point while they are in the study, they will exit the study protocol and receive standard treatment for hip dysplasia as medically indicated.

Basic demographics initially (gender, race/ethnicity, age of the mother), birth presentation (normal or breach), multiple birth, the number of births that the mother has had, family history of hip dysplasia, gestational age, alpha angle and percent coverage as defined above (measured by three independent observers) will be collected at the initial exam. At each follow up exam the following data will be collected; date of exam, gestational age, corrected age, alpha angle, percent coverage and any notes about the exam. In addition, contact information will be collected so that follow up visits can be scheduled. All data will be entered into REDCap, UCSF's HIPAA compliant data entry site.

ELIGIBILITY:
Inclusion Criteria:

* newborns born at CRMC (term newborns and pre-mature newborns over 32 weeks gestational age.
* newborns in NICU
* newborns on postpartum floor
* single birth
* multiple births
* normal presentation
* breach presentation

Exclusion Criteria:

* known neuromuscular or genetic condition predisposing infant to hip dysplasia (i.e. Spina Bifida, Cerebral Palsy),
* inability to follow up (i.e. doesn't live in surrounding area),
* frankly dislocated hips that require immediate treatment,
* any medical condition precluding safe hip ultrasound.

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Convenience sample of of newborns that are born at Community Regional Medical Center (CRMC).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Alpha Angle in degrees | Measured weekly from birth to 6 weeks corrected age
  The angle between the roof of the acetabulum and the lateral iliac wing and indicates,morphology of the acetabulum.
Percent Coverage | Measured weekly from birth to 6 weeks corrected age
  Percent coverage of the femoral head in the acetabulum

CONTACTS AND LOCATIONS:
Overall Officials: John Wiemann, MD, Principal Investigator — UCSF - Fresno
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No